CLINICAL TRIAL: NCT01929135
Title: Short-term Effect of 2% Atorvastatin Dentifrice as an Adjunct to Periodontal Therapy: A Randomized Double-blind Clinical Trial.
Brief Title: Short-term Effect of 2% Atorvastatin Dentifrice in Periodontal Status.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Corporación de Fomento de la Producción, Chile (Unknown)
Responsible Party: Principal Investigator, Dr. David Rosenberg, Associate Professor of the Faculty of Dentistry, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORFO-13IDL1-18270
Record Dates: First submitted 2013-08-18; First posted 2013-08-27 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Periodontitis
Keywords: Periodontal Disease; Chronic Periodontitis; Atorvastatin; Statins; Hydroxymethylglutaryl-coenzyme A Reductase Inhibitors; Dentifrice
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medicated 2% atorvastatin dentifrice (Experimental): A group of 19 patients received non surgical periodontal therapy accompanied by instruction for oral hygiene, using a medicated 2% atorvastatin dentifrice 2 times a day for two minutes each time, for 30 days.
  Interventions: Drug: Medicated 2% atorvastatin dentifrice
- Non-medicated dentifrice (Placebo Comparator): A group of 19 patients received non surgical periodontal therapy accompanied by instruction for oral hygiene, using a non-medicated dentifrice as placebo 2 times a day for two minutes each time, for 30 days.
  Interventions: Drug: Non-medicated dentifrice

INTERVENTIONS:
Drug: Medicated 2% atorvastatin dentifrice — Non surgical periodontal therapy accompanied by medicated 2% atorvastatin dentifrice (20 mg per ml) 2 times a day for two minutes each time, for 30
  Other Names: medicated dentifrice with atorvastatin
  Arms: Medicated 2% atorvastatin dentifrice
Drug: Non-medicated dentifrice — Non surgical periodontal therapy accompanied by non medicated dentifrice 2 times a day for two minutes each time, for 30 days.
  Other Names: Placebo dentifrice
  Arms: Non-medicated dentifrice

SUMMARY:
Periodontal disease (PD) is an inflammatory, infectious and destructive condition of the tissues surrounding the teeth. However, even if bacteria are required to initiate periodontal disease, the immune response is responsible for most of the destruction of the periodontal tissues. Statins may be used to control the immune response to periodontal pathogens, a factor that has not yet been managed clinically and even less massively.

Recently it has been reported the pharmacological effectiveness of topically used statins. For periodontal disease, at least four well conducted clinical trials have been published using a topically statin formula for pocket irrigation in adult populations with chronic periodontal disease, observing surprising clinical results in all of them (with clinical and statistical significance) and no adverse reactions.

The purpose of the present study is asses the effectiveness of a medicated 2% atorvastatin dentifrice, as complement to non-surgical conventional periodontal treatment. Clinical examination will be made at the beginning and after one month of treatment.

DETAILED DESCRIPTION:
An medicated 2% atorvastatin dentifrice (2 mg x every 0.1 ml of dentifrice) will be prepared for dental brushing. It will be used as a base a fluoride dentifrice, to which will be added atorvastatin in the prescribed amount. Medicated prototypes and placebos will be dosed in 5 ml syringes indicating each 0.5 ml measures to facilitate dispensing the product and ensure proper use. Thus, each syringe will be for 10 doses of toothpaste (10 brushings). 6 syringes will be provided to each patient, so that they have enough for a month of treatment, during which they will have to brush 2 times a day.

Sample size:

A clinical trial with two parallel groups (1:1) will be conducted, where there will be 2 groups of 19 patients each. The estimated sample size was based on the difference in attachment level achieved in the study Goodson et al (Goodson, Haffajee, Socransky, Kent, Teles, Hasturk, Bogren, Van Dyke, Wennstrom, Lindhe. Control of periodontal infections: A randomized controlled trial I. The primary outcome attachment gain and pocket depth reduction at Treated sites. J Clin Periodontol 2012, 39: 526-536), with a power of 90%, a significance level of 0.05 two-tailed.

Treatments and protocols:

Patients will be treated at the Department of Periodontology of Health Care Center, Universidad de Los Andes in San Bernardo, Santiago, Chile.

The two groups will undergo non-surgical periodontal therapy consisting of scaling and root planning of all tooth groups.

Therapy will be supplemented with oral hygiene instruction, indicating patients to brush with the dentifrice that will be provided, 2 times a day for two minutes each time. Then they will be told to spit the dentifrice excesses during 30 seconds, but not to rinse their teeth, or consume liquids or solid foods for at least 30 minutes. A group of 19 patients will receive the medicated 2%atorvastatin dentifrice while the other group of 19 patients will receive dentifrice without the drug to act as a placebo.

The record of the application of statins will be done by a professor at the Faculty of Dentistry, before periodontal clinical evaluation, in order not to influence the researcher.

The allocation to each group will be random and there will be a sequence concealment.

Analysis Plan:

Continuous variables will be described by measures of central tendency and dispersion. Dichotomous variables will be tabulated and described by absolute frequencies and percentages according to each group. The delta of the outcome variables will be calculated as the difference between measurements before and after intervention. Multiple linear regression models will be used to compare the deltas of outcome variables after adjusting for gender, diabetes and tobacco use. A p value of <0.05 is considered statistically significant. The analysis will be performed with Stata software (version 12; Stata Corporation, Lakeway Drive, College Station, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study will be those fully agreeing to participate by signing an informed consent, which has been submitted to and approved, together with the study protocol by the Ethics Committee of the Faculty of Dentistry of Universidad de Los Andes.
* The target population consists of 38 adult patients who consult the Service of Periodontology at the Universidad de Los Andes.
* The eligible population are those that meet the following criteria:

  1. more than 35 years of age.
  2. with at least 14 natural teeth in mouth (excluding third molars).
  3. have some degree of periodontal disease.

Exclusion Criteria:

* Will be excluded those who:

  1. Relate migration plans.
  2. Presence of limiting disease for the understanding and execution of the study or are hospitalized.
  3. Received periodontal treatment in the last year.
  4. Completed antibiotic therapy or Non Steroidal Anti-inflammatory Drugs (NSAIDs) in the last two weeks.
  5. Are using calcium channel blockers, phenytoin, cyclosporine or any associated drug that may affect gingival tissue.
  6. Have autoimmune pathology.
  7. Require antibiotic prophylaxis for periodontal treatment.
  8. Patients requiring treatment with NSAIDs for postoperative pain control after the procedure done.
  9. Patients on statin therapy for dyslipidemia.
  10. Pregnant patients.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Rosenberg, DDS, MDS, Principal Investigator — Universidad de Los Andes
Locations (2):
- Chile (2):
  - Centro de Salud Universidad de los Andes, San Bernardo, Santiago, Santiago Metropolitan
  - CIBRO Universidad de los Andes, Santiago, Santiago Metropolitan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigation was conducted at the Department of Periodontology of Universidad de Los Andes.
  Patients were enrolled in the study between June 2013 and August 2013, derived from the Health Care Center, Universidad de los Andes (San Bernardo, Santiago, Chile).
Groups:
- Atorvastatin Group: A group of 19 patients received non surgical periodontal therapy accompanied by instruction for oral hygiene, using a medicated 2% atorvastatin dentifrice 2 times a day for two minutes each time for a period of 30 days..
- Placebo Group: A group of 19 patients received non surgical periodontal therapy accompanied by instruction for oral hygiene, using a non-medicated dentifrice as placebo 2 times a day for two minutes each time, for 30 days.
Period: Overall Study
Arm/Group | Atorvastatin Group | Placebo Group
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin Group | Placebo Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.39 (9.07) | 45.72 (9.08) | 45.56 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 4 | 7 | 11
Diabetic [Number; unit: participants]
  diabetic patients | 3 | 1 | 4
  non-diabetic patients | 15 | 17 | 32
Smokers [Number; unit: participants]
  smokers patients | 5 | 11 | 16
  non-smokers patients | 13 | 7 | 20
Probing depth [Mean (Standard Deviation); unit: millimeters] — Probing depth (PD) was defined as the distance from the gingival margin to the base of clinical pocket, was measured as the distance between the base of the clinical pocket and the cement-enamel junction (CEJ) using University of North Carolina no. 15 color-coded periodontal probe, Hu-Friedy.
  millimeters | 3.74 (0.87) | 2.80 (0.86) | 3.27 (0.98)
Clinical attachment level [Mean (Standard Deviation); unit: millimeters] — Clinical attachment level (CAL) was measured as the distance between the base of the clinical pocket and the cement-enamel junction (CEJ) using a University of North Carolina no. 15 color-coded periodontal probe, Hu-Friedy.
  millimeters | 3.73 (1.52) | 2.52 (0.90) | 3.12 (1.38)
Bleeding on probing [Mean (Standard Deviation); unit: Percentage of probed sites with BOP] — Bleeding on probing (BOP) was determined by assigning with positive sign (+) when presence of bleeding on probing in buccal and / or palatal of an examined tooth; and with a negative sign (-) when not bleeding. Then the positive signs were summed and divided by the number of examined sites obtaining a percent. Each tooth was probed at 6 sites: mesiobuccal, mediobuccal, distobuccal, mesiolingual, mediolingual, distolingual.
  Percentage of probed sites with BOP | 77.86 (18.12) | 53.47 (17.77) | 65.67 (21.59)
Recession [Mean (Standard Deviation); unit: millimeters] — Recession was defined as the distance from gingival margin to cemento-enamel junction (CEJ) registered as a negative value when gingival margin extends under CEJ or positive value in case of the gingival margin extends upper CEJ. Each tooth was measured at 6 sites: mesiobuccal, mediobuccal, distobuccal, mesiolingual, mediolingual, distolingual. The mean of all examined sites was calculated in each patient.
  millimeters | 0.01 (1.14) | 0.28 (0.94) | 0.14 (1.04)
Oral hygienic index [Mean (Standard Deviation); unit: percent of surface without plaque] — The Oral hygienic index was evaluated recording the presence and absence of plaque on surfaces examined (mesiobuccal, mediobuccal, distobuccal, mesiolingual/palatal, mediolingual/palatal, distolingual/palatal), then the percentage of surface without plaque was calculated.
  percent of surface without plaque | 7.32 (16.85) | 12.88 (18.01) | 10.10 (17.42)
Gingival index [Mean (Standard Deviation); unit: score on a scale] — Determined as score assigned to each site evaluated respect to clinical criteria as followed:
  Score Criteria 0: No inflammation
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  Then was calculated a score for each sextant summed the score and divided by the number of examined sites. Later was summed each sextant score and divided by sextant evaluated.
  score on a scale | 1.95 (0.31) | 1.54 (0.21) | 1.74 (0.33)
Periodontal inflamed surface area (PISA) [Mean (Standard Deviation); unit: square millimeters] — Periodontal Inflamed Surface Area (PISA) was calculated using formulas with data of CAL, Gingival Recession and BOP obtaining surface area of bleeding pocket epithelium in square millimetres. A freely downloadable spreadsheet available was used to calculate PISA (http://www.parsprototo.info)
  square millimeters | 1093.18 (435.96) | 814.82 (488.54) | 954 (477.67)

OUTCOME MEASURES:

1. Primary Outcome: Change in Periodontal Inflammation Surface Area (PISA)
Description: PISA will be computed through an Excel spreadsheet, using data of clinical attachment level, gingival recession and bleeding on probing.
  Change in PISA: baseline measure minus 1 month later measure.
Time Frame: baseline and 1 month later of intervention
Measure: Mean (Standard Deviation); unit: square millimeters
Groups:
- Atorvastatin Toothpaste: A group of 19 patients will receive the Atorvastatin 2% toothpaste. Therapy will be supplemented with oral hygiene instruction, indicating patients to brush with the toothpaste 2 times a day for two minutes each time for a period of 30 days.
  Atorvastatin: Toothpaste with Atorvastatin 2% (20 mg per ml), brushing 1 minute 2 time a day, for 30 days.
- Non Medicated Gel Toothpaste: A group of 19 patients will receive a toothpaste without the drug to act as a placebo.Therapy will be supplemented with oral hygiene instruction, indicating patients to brush with the toothpaste that will be provided, 2 times a day for two minutes each time, for 30 days.
  Non medicated gel toothpaste: Normal gel toothpaste used as placebo, brushing 1 minute 2 time a day, for 30 days.
Arm/Group | Atorvastatin Toothpaste | Non Medicated Gel Toothpaste
Number analyzed (Participants) | 18 | 18
square millimeters | 638.16 (398.74) | 288.72 (168.20)

2. Secondary Outcome: Change in Mean Pocket Depth (PD)
Description: The PD will be defined as the distance from the free gingival margin to the bottom of the pocket. For each tooth will be conducted periodontal probing at 6 sites (mesiobuccal, mediobuccal, distobuccal, mesiolingual / palatal, mediolingual / palatal, distolingual/ palatal).
  Change in mean PD: baseline measure minus 1 month later measure.
Time Frame: baseline and 1 month later
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Atorvastatin Toothpaste | Non Medicated Gel Toothpaste
Number analyzed (Participants) | 18 | 18
millimeters | 1.29 (0.45) | 0.70 (0.53)

3. Secondary Outcome: Change in Clinical Attachment Level (CAL)
Description: The Clinical Attachment Level (CAL) is defined as the distance from the cement-enamel junction to the fornix of the pocket. For each tooth will be performed periodontal probing at 6 sites (mesiobuccal, mediobuccal, distobuccal mesiolingual / palatal mediolingual / distolingual palatal / lingual).
  Change in CAL: baseline measure minus 1 month later measure.
Time Frame: baseline and 1 month after intervention
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Atorvastatin Toothpaste | Non Medicated Gel Toothpaste
Number analyzed (Participants) | 18 | 18
millimeters | 0.89 (0.33) | 0.49 (0.31)

4. Secondary Outcome: Change in Bleeding on Probing Index (BOP)
Description: The bleeding on probing index (BOP) will be determined by assigning + to the presence of bleeding on vestibular / palatine probing of the tooth examined and with a sign - the abscence. Later the + signs will be summed and divided by the number of sites examined.
  Change in BOP: baseline measure minus 1 month later measure.
Time Frame: baseline and 1 month after intervention
Measure: Mean (Standard Deviation); unit: percentage of BOP
Arm/Group | Atorvastatin Toothpaste | Non Medicated Gel Toothpaste
Number analyzed (Participants) | 18 | 18
percentage of BOP | 64.42 (18.08) | 28.56 (15.56)

5. Secondary Outcome: Change in Gingival Index
Description: Determined as score assigned to each site evaluated respect to clinical criteria as followed:
  Score Criteria:
  0. No inflammation
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  Then was calculated a score for each sextant summed the score and divided by the number of examined sites. Later was summed each sextant score and divided by sextant evaluated.
  The change was calculated as baseline measure minus 1 month later measure.
Time Frame: baseline and 1 month after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Atorvastatin Group: A group of 19 patients will receive the Atorvastatin 2% toothpaste. Therapy will be supplemented with oral hygiene instruction, indicating patients to brush with the toothpaste 2 times a day for two minutes each time for a period of 30 days.
  Atorvastatin: Toothpaste with Atorvastatin 2% (20 mg per ml), brushing 1 minute 2 time a day, for 30 days.
Arm/Group | Atorvastatin Group | Placebo Group
Number analyzed (Participants) | 18 | 18
score on a scale | 1.04 (0.54) | 0.54 (0.42)

ADVERSE EVENTS:
Time Frame: one month
Description: After treatment, patients were telephoned every week, to consult for any reaction to dentifrice
Groups:
- Atorvastatin Group: A group of 19 patients received Non-surgical periodontal treatment (NSPT) plus medicated 2% atorvastatin dentifrice. Therapy was supplemented with oral hygiene instruction, indicating patients to brush with the dentifrice 2 times a day for two minutes each time for a period of 30 days.
  Atorvastatin dentifrice: fluoride dentifrice with 2% Atorvastatin (20 mg per ml).
- Placebo Group: A group of 19 patients received Non-surgical periodontal treatment (NSPT) plus placebo dentifrice.Therapy was supplemented with oral hygiene instruction, indicating patients to brush with dentifrice 2 times a day for two minutes each time, for 30 days.
  Non medicated dentifrice: fluoride dentifrice.
Arm/Group | Atorvastatin Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No